CLINICAL TRIAL: NCT04192110
Title: Association of Diuretics With Change in Extracellular Volume, Natriuretic Peptides, Symptoms, and Cardiovascular Outcomes in CKD
Acronym: DOCK
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: The project has ended prior to beginning.
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NEPH-025-19S; 1IK2CX002030-01 (NIH)
Record Dates: First submitted 2019-12-06; First posted 2019-12-10 (Actual); Last update posted 2021-12-09 (Actual); Status verified 2021-12

CONDITIONS: Chronic Kidney Disease
Keywords: Chronic kidney disease; Diuretics; Volume overload; Natriuretic peptides; Bioimpedance spectroscopy; Cardiovascular disease
MeSH Terms: conditions — Renal Insufficiency, Chronic; Edema; Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: Single group open label initiation or dose increase of loop or thiazide-type diuretics
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Diuretic initiation or augmentation (Experimental): Participants will either initiate or increase the dose of a loop or thiazide-type diuretic
  Interventions: Drug: Diuretic initiation or augmentation

INTERVENTIONS:
Drug: Diuretic initiation or augmentation — The participant's blood pressure medication regimen will then be altered to initiate a thiazide-type (hydrochlorothiazide or chlorthalidone) or loop diuretic (furosemide, bumetanide, or torsemide) in those not already prescribed a diuretic, or to increase the dose if one is already prescribed

SUMMARY:
Almost 15% of Americans have chronic kidney disease (CKD), with an even higher rate in Veterans due to common risk factors such as high blood pressure and diabetes. People with CKD have a high risk of cardiovascular (CV) diseases, such as heart attacks, heart failure, and strokes. Extra fluid in the body, called volume overload, may lead to CV disease in people with CKD. It is unknown if volume overload develops in the earliest stages of CKD, when treating it with common, inexpensive medicines called diuretics may improve long-term CV outcomes. This study will lay important groundwork to answer this question in Veterans with early CKD by comparing two ways to measure volume overload and studying the change in common symptoms like fatigue and short-term CV function after treatment with diuretic medicines.

DETAILED DESCRIPTION:
The investigators previously showed that brain natriuretic peptide (BNP) and N-terminal-pro-BNP (NT-pro-BNP), measures of ventricular stretch, are associated with death and cardiovascular (CV) outcomes in chronic kidney disease (CKD) stages 1-3 patients, and the investigators' preliminary pilot results suggest that these natriuretic peptides may correlate with objective measures of excess extracellular volume (ECV) and with symptoms common in CKD. The overarching objective is to determine if initiation of diuretic treatment or increase in dose is associated with changes in BNP and NT-pro-BNP, patient-reported symptom burden, and short-term hemodynamic parameters in patients with CKD stages 1-3 and elevated blood pressure, and whether these changes correlate with changes in ECV. The central hypothesis is that the change in ECV after starting or increasing diuretics in Veterans with stages 1-3 CKD is associated with changes in 1) natriuretic peptides, 2) patient-level factors, and 3) CV physiology.

The investigators will compare the changes in natriuretic peptides, symptoms, and CV parameters with the change in ECV after diuretic initiation or dose increase. The primary aim is to determine if initiation of diuretic treatment or increase in diuretic dose is associated with changes in natriuretic peptides. Secondary aims are to determine the effect of diuretic change on patient-reported symptom burden, and CV physiology.

This clinical trial will include 46 outpatients with CKD stages 1-3 and blood pressure >140/90 mmHg. At the first visit, I will initiate or increase the dose of a thiazide or loop diuretic. Study measures other than echocardiogram will be repeated 4 weeks after the intervention to determine changes in these parameters. ECV will be measured by whole-body multifrequency bioimpedance spectroscopy (BIS), which is a validated, non-invasive, painless measure of ECV. Plasma BNP and NT-pro-BNP will be measured, and patient-reported fatigue, depression, and quality of life will be quantified using validated questionnaires. Hemodynamic parameters include blood pressure, pulse pressure, total peripheral resistance index (TPRI), and cardiac index measured by Non-Invasive Cardiac Output Monitoring. A transthoracic echocardiogram will measure left ventricular mass index, valvular disease, and diastolic dysfunction.

Variables will be compared within participants between baseline and Visit 2 using paired Wilcoxon Signed Rank tests or paired Student's t tests, depending on variable distributions. Correlations between change in ECV/total body weight and all continuous outcome measures will be analyzed using Spearman or Pearson correlations, applying appropriate transformations. Linear regression analysis will control for clinically relevant variables. The relationship between ECV/total body weight and natriuretic peptides from both visits will be evaluated using a mixed effects model to account for the change in these measures between baseline and Visit 2.

This study is minimal risk to human subjects. Participants may benefit from improved control of their blood pressure. The knowledge to be gained may also benefit others in the future.

ELIGIBILITY:
Inclusion Criteria:

* The presence of CKD stages 1, 2, or 3, as defined below by National Kidney Foundation guidelines, for a period of at least 3 months.

  * Stage 1: eGFR 90 mL/min/1.73 m2 and spot urine albumin-to-creatinine ratio 30 mg/g.
  * Stage 2: eGFR 60-89 mL/min/1.73 m2 and spot urine albumin-to-creatinine ratio 30 mg/g.
  * Stage 3: eGFR 30-59 mL/min/1.73 m2.
* Measured blood pressure either >140 mmHg systolic or >90 mmHg diastolic at the two most recent clinic visits.

  * Rationale: The investigators' unpublished preliminary data show that blood pressure correlates with both BNP and NT-pro-BNP more strongly in those with CKD than those without CKD. Thus, selecting hypertensive individuals is more likely to identify those with elevated natriuretic peptides in the CKD group.
  * Furthermore, starting or increasing a diuretic medication is part of standard of care to treat blood pressures >140/90 mmHg, so the study intervention will be consistent with appropriate care for the Veteran and avoid hypotension.
* Able to understand and sign informed consent after the nature of the study has been fully explained.

Exclusion Criteria:

* Unable to understand or provide informed consent.
* Unwilling or unable to participate in the protocol or comply with any of its components.
* CKD stages 4-5, defined as eGFR <30 mL/min/1.73 m2.
* Receiving chronic hemodialysis or peritoneal dialysis.
* Recipient of a kidney transplant.
* Serum potassium <3.5 mg/dL at baseline.
* Known left ventricular ejection fraction <40% on visual estimate based on chart review of available echocardiogram data.
* Known hepatic cirrhosis.
* Major limb amputation.
* Known pregnancy.
* Presence of a pacemaker or defibrillator.
* Presence of metal prostheses.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-08-11 (Actual); Primary Completion 2020-08-11 (Actual); Study Completion 2020-08-11 (Actual)

PRIMARY OUTCOMES:
NT-pro-BNP | 4 weeks
  Change from baseline to 4 weeks in NT-pro-BNP
Total peripheral resistance index | 4 weeks
  The change from baseline to 4 weeks in total peripheral resistance index will be measured using Non-Invasive Cardiac Output Monitoring (Cheetah)

SECONDARY OUTCOMES:
BNP | 4 weeks
  Change from baseline to 4 weeks in BNP
Fatigue | 4 weeks
  The change in fatigue from baseline to 4 weeks, measured by the Functional Assessment of Chronic Illness Therapy - Fatigue, a validated measure of patient-reported fatigue
Depression | 4 weeks
  The change in depressive symptoms from baseline to 4 weeks, measured by the Quick Inventory of Depressive Symptomatology, a validated measure of patient-reported depression
Quality of Life - Kidney Disease Quality of Life (KDQOL) | 4 weeks
  The change in quality of life from baseline to 4 weeks, measured by the KDQOL, a validated measure of patient-reported quality of life
Hospitalizations | 6 months
  Hospitalizations as quantified by review of the medical record and telephone contact with the participant
Systolic blood pressure | 4 weeks
  The change in systolic blood pressure from baseline to 4 weeks
Diastolic blood pressure | 4 weeks
  The change in diastolic blood pressure from baseline to 4 weeks
Mean arterial blood pressure | 4 weeks
  The change in mean arterial blood pressure from baseline to 4 weeks
Pulse pressure | 4 weeks
  The change in pulse pressure from baseline to 4 weeks
Cardiac index | 4 weeks
  The change from baseline to 4 weeks in cardiac index will be measured using Non-Invasive Cardiac Output Monitoring (Cheetah)

OTHER OUTCOMES:
Evolume | 4 weeks
  The change in extracellular fluid volume from baseline to 4 weeks, measured by multifrequency bioimpedance spectroscopy and normalized to total body weight

CONTACTS AND LOCATIONS:
Overall Officials: Lucile P Gregg, MD, Principal Investigator — VA North Texas Health Care System Dallas VA Medical Center, Dallas, TX
Locations (1):
- VA North Texas Health Care System Dallas VA Medical Center, Dallas, TX, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No